CLINICAL TRIAL: NCT03152942
Title: A Randomised Controlled Feasibility Study of the Tolerability of the Combination of Progesterone and Aminophylline for the Prevention of Preterm Labour
Brief Title: Progesterone and Aminophylline for the Prevention of Preterm Labour
Acronym: PROGRAM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Stephens Aids Trust (Other)
Collaborators: Action Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSAT068
Record Dates: First submitted 2016-07-03; First posted 2017-05-15 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2017-10

CONDITIONS: Premature Obstetric Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Progesterone; Aminophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Progesterone alone (Experimental): Progesterone 400 mg once daily until 34 weeks.
  Interventions: Drug: Progesterone
- Progesterone and aminophylline. (Active Comparator): Progesterone 400 mg and aminophylline 225 mg once daily until 34 weeks.
  Interventions: Drug: Progesterone; Drug: Aminophylline

INTERVENTIONS:
Drug: Progesterone — Progesterone 400mg to be administered once daily for 34 weeks in the patients randomised to receive progesterone alone
  Other Names: Cyclogest
Drug: Aminophylline — Patients randomised to the combination arm to be administered aminophylline 225 mg to be taken once at night for 1 week and then if tolerated increased to 225 mg twice daily Progesterone 400mg to be administered once daily for 34 weeks.
  Other Names: Phyllocontin® Continus®
  Arms: Progesterone and aminophylline.

SUMMARY:
The aim of this study is to investigate whether the combination of aminophylline and Progesterone (P4) is acceptable to women at high-risk of Pre-term labour (PTL). If this proves to be the case, a larger double blind, randomised controlled trial will be conducted to test the hypothesis that the combination of P4 and aminophylline reduces the risk of PTL more effectively than P4 alone.

The study is a randomised study where participants will be either administered a combination of aminophylline and Progesterone (P4) or Progesterone (P4) alone.As the study is open label, the participants and the study doctor will know which study medications the participant is taking at all times during the study.

DETAILED DESCRIPTION:
Name of Investigational Product: Cyclogest® 400 mg, Phyllocontin® Continus®

Name of active ingredients:Progesterone PhEur 400 mg, Aminophylline hydrate 225 mg

Phase of study: Phase I

Primary Objectives:

1. To assess how many women at high risk of Preterm Labour (PTL) withdraw from the combination therapy of Progesterone (P4) and aminophylline due to side effects in comparison to P4 alone.

Secondary Objectives:

1. The effect on the maternal immune system.
2. The impact on preterm delivery and episodes of threatened PTL.
3. The number of women who deliver before 34 weeks.

Methodology:

This randomised controlled feasibility study will establish the viability of conducting a multicentre randomised controlled study to definitively test the effects of the combination of Progesterone (P4) and aminophylline against P4 alone.

Participants (n=70) will be randomised into one of two groups. One group will receive P4 alone while the second group will receive a combination of P4 and aminophylline. Following randomisation to P4 alone or in combination with aminophylline, participants will be given a prescription to be taken to the pharmacy.

All participants will be given a prescription for P4 400 mg to be inserted into the vagina at bedtime until 34 weeks.

Participants randomised to the combined arm will also be given a prescription for aminophylline 225 mg to be taken once at night for 1 week and then if tolerated increased to 225 mg twice daily.

Subjects will attend the unit for 34 weeks for clinical review and safety monitoring. Treatment will be continued until 34 weeks of gestation or until preterm delivery (whichever occurs first).

During the safety visits, flow cytometry will be used to determine inflammatory cell numbers and their activation status in cervical and blood samples.

Cervico-vaginal fluid and peripheral blood plasma will also be stored at - 80oC until multiplex analysis of cytokine and chemokine content.

Summary of eligibility criteria:

* Obstetric history: previous mid-trimester loss and preterm delivery
* Short cervical length (≤ 25 mm) on ultrasound at 13-20+0 weeks gestation, with or without a cervical suture and with or without a positive fetal fibronectin
* Women must be aged 18 years or older

Primary Endpoint:

1. The number of women maintained on the combination therapy P4 and aminophylline arm and the P4 alone alrm up to 34 weeks of treatment. A positive outcome would be seeing 80% or more women maintained on therapy.

Secondary Endpoint:

1. The effects on the maternal immune system.
2. The number of women who deliver before the end of the study (34 weeks).
3. The impact on preterm delivery and episodes of threatened PTL.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women between 13 and 20 weeks of gestation.
2. Singleton pregnancy.
3. Intact fetal membranes at the time of recruitment.
4. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements.
5. Obstetric history: previous mid-trimester loss (14 - 26 weeks) and preterm delivery (< 37 weeks).
6. Women with a history of indicated cervical suture.
7. Short cervical length (≤ 25 mm) on ultrasound at 13-20+0 weeks gestation, with or without a cervical suture and with or without a positive fetal fibronectin.
8. Women must be aged 18 years or older.

Exclusion Criteria:

1. Known sensitivity, contraindication or intolerance to P4 (History of liver tumours, severe liver impairment, genital or breast cancer, severe arterial disease, undiagnosed vaginal bleeding, acute porphyria, history during pregnancy of idiopathic jaundice, severe pruritus or pemphigoid gestations)
2. Known sensitivity, contraindication or intolerance to aminophylline (hypokalaemia, pre-existing cardiac arrhythmias, epilepsy, hyperparathyroidism, peptic ulcer disease)
3. Suspected or proven rupture of the fetal membranes at the time of recruitment.
4. Prescription or ingestion of medications known to interact with P4 (e.g Bromocriptine, carbamazepine, diazepam, lorazepam and temazepam, insulin).
5. Aminophylline plasma concentrations can be increased in the presence of: acyclovir, calcium channel blockers, cimetidine, erythromycin, clarithromycin, corticosteroids and benzodiazepine, carbamazepine, beta-sympathomimetics.
6. Evidence of maternal infection or sepsis (maternal temperature ≥37.5C, increased inflammatory markers - WBC, CRP).
7. Multiple pregnancy.
8. Known significant congenital structural or chromosomal fetal anomaly.
9. Maternal pathologies in which preterm termination of pregnancy is required.
10. Pre-eclampsia or severe hypertension.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
To assess number of women at high risk of Preterm Labour (PTL) withdraw from the combination therapy of Progesterone (P4) and aminophylline due to side effects, in comparison to P4 alone. | 34 weeks
  Tolerability will be assessed by the number of participants who withdraw from the study due to severe adverse side effects at each safety visit (14, 16, 18, 22, 26, 30 and 34 weeks of pregnancy).

SECONDARY OUTCOMES:
To assess the effect on the maternal immune system. | 34 weeks
  By studying cervicovaginal swabs taken every 4 weeks, blood tests, and measuring levels of cytokine and chemokine inflammatory profile.
The impact on preterm delivery and episodes of threatened Preterm Labour | 34 weeks
  This will be measured by number of preterm deliveries and reported side effects between the two groups on combination and mono therapy.
The number of women who deliver before 34 weeks. | 34 weeks
  Measuring the number of patients who deliver before 34 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Johnson, Professor, Principal Investigator — Chelsea and Westminster Hospital
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh N, Shah NM, Sooranna G, Bourke M, Yulia A, Battersby C, Tribe RM, Johnson MR. A randomised feasibility tolerability study of aminophylline for the prevention of preterm labour. BMC Pregnancy Childbirth. 2025 Mar 27;25(1):357. doi: 10.1186/s12884-025-07488-1. PMID 40148792